CLINICAL TRIAL: NCT05059366
Title: Improvement of Manual Ventilation Efficacy With Ventilation Grip Device: A Manikin Study
Brief Title: Manual Ventilation Efficacy With MVG Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Alecia Stein, Assistant Professor of Clinical, University of Miami
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 20200039
Record Dates: First submitted 2021-09-03; First posted 2021-09-28 (Actual); Results first posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Ventilator Lung
Keywords: Manual Ventilation Grip Device

STUDY DESIGN:
Intervention Model Description: The study is a repeated-measures cross over design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Expert participants randomized to MVG followed by 2VE (Experimental): Expert participants (Anesthesiology residents and attendings with at least 2 or more years of clinical experience) randomized to perform the ventilation on a manikin using the Manual ventilation grip device (MVG) first followed by the standard 2VE technique alone.
  Interventions: Device: Manual Ventilation Grip Device; Other: 2VE
- Expert participants randomized to 2VE followed by MVG (Experimental): Expert participants (Anesthesiology residents and attendings with at least 2 or more years of clinical experience) randomized to perform the ventilation on a manikin using the standard technique (2VE) alone first followed by Manual ventilation grip device (MVG).
  Interventions: Device: Manual Ventilation Grip Device; Other: 2VE
- Novice participants randomized to MVG followed by 2VE (Experimental): Novice participants (Current medical students or residents with no prior experience in hand mask ventilation techniques) first followed by the standard technique (2VE) alone
  Interventions: Device: Manual Ventilation Grip Device; Other: 2VE
- Novice participants randomized to 2VE followed by MVG (Experimental): Novice participants (Current medical students or residents with no prior experience in hand mask ventilation techniques) randomized to perform the ventilation on a manikin using the standard technique (2VE) alone first followed by Manual ventilation grip device (MVG)
  Interventions: Device: Manual Ventilation Grip Device; Other: 2VE

INTERVENTIONS:
Device: Manual Ventilation Grip Device — Manual Ventilation Grip Device is an add-on device placed on a standard valve mask to assist ventilation.
Other: 2VE — the standard 2VE technique for ventilation

SUMMARY:
The purpose of this research is to investigate the efficacy of the newly designed ventilation grip device (MVG device).

ELIGIBILITY:
Inclusion Criteria:

1. Current medical students, Post Graduate Year 1 (PGY1) residents or residents from other specialties with no prior experience in hand mask ventilation techniques or anesthesiology residents and attendings with at least 2 or more years of clinical experience

Exclusion Criteria:

1. Refusal to participate in the study.
2. Medical students with prior experience in hand mask ventilation techniques (i.e. experiences in previous careers such as nursing or Emergency Medical Technician (EMT) professions)
3. Any physical inability to adequately perform ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alecia Stein, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Expert Participants Randomized to MVG Followed by 2VE | Expert Participants Randomized to 2VE Followed by MVG | Novice Participants Randomized to MVG Followed by 2VE | Novice Participants Randomized to 2VE Followed by MVG
Started | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Experts Group: Anesthesiology residents and attendings with at least 2 or more years of clinical experience conducting both the Manual ventilation grip device (MVG) and the standard 2VE technique.
- Novices Group: Current medical students or residents with no prior experience in hand mask ventilation techniques conducting both the Manual ventilation grip device (MVG) and the standard 2VE technique.
- Total: Total of all reporting groups
Arm/Group | Experts Group | Novices Group | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 32
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 9 | 8 | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Tidal Volume
Description: As measured using the ventilator machine in milliliters
Time Frame: Day 1
Population: 3 participants in the experts group were excluded due to unresolvable set-up obstacles
Measure: Mean (Standard Error); unit: mL
Arm/Group | Experts Group | Novices Group
Number analyzed (Participants) | 13 | 16
mL
  MVG technique | 502.030 (11.372) | 492.508 (10.220)
  2VE technique | 478.889 (12.462) | 481.533 (11.200)

2. Secondary Outcome: Fatigue as Measured by NASA-TLX Questionnaire
Description: NASA Task Load Index (TLX) questionnaire has a total overall workload score ranging from 0 and 126 with the higher score indicating greater demand.
Time Frame: Day 1
Population: 3 participants in the experts group were excluded due to unresolvable set-up obstacles
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Experts Group | Novices Group
Number analyzed (Participants) | 13 | 16
score on a scale
  MVG technique | 33.92 (5.23) | 53.69 (6.74)
  2VE technique | 42.54 (5.24) | 63.69 (6.28)

3. Secondary Outcome: Fatigue as Measured by SOFI Questionnaire
Description: Swedish Occupational Fatigue Inventory (SOFI) questionnaire has a total score ranging from 0 to 120 with the higher score indicating greater fatigue
Time Frame: Day 1
Population: 3 participants in the experts group were excluded due to unresolvable set-up obstacles
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Experts Group | Novices Group
Number analyzed (Participants) | 13 | 16
score on a scale
  MVG technique | 13.08 (3.32) | 17.13 (2.97)
  2VE technique | 16.38 (3.13) | 23.28 (2.74)

ADVERSE EVENTS:
Time Frame: 1 day
Description: The study is a cross-over design. All participants received both the MVG and 2VE intervention.
Groups:
- Manual Ventilation Grip Device (MVG): Manual Ventilation Grip Device is an add-on device placed on a standard valve mask to assist ventilation.
- Standard Technique (2VE): The standard 2VE technique for ventilation
Arm/Group | Manual Ventilation Grip Device (MVG) | Standard Technique (2VE)
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-21): https://cdn.clinicaltrials.gov/large-docs/66/NCT05059366/Prot_SAP_000.pdf